CLINICAL TRIAL: NCT02150538
Title: BiventRicular Pacing in prolongEd Atrio-Ventricular intervaL: the REAL-CRT Study
Acronym: REAL-CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gianluca Botto (Other)
Responsible Party: Sponsor-Investigator, Gianluca Botto, Head of Electrophysiology Unit, S. Anna Hospital
Organization: S. Anna Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Parere Unico 86/13
Record Dates: First submitted 2014-04-15; First posted 2014-05-30 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: First Degree Atrioventricular Block
Keywords: Cardiac Resynchronization therapy; Minimized Right ventricular pacing; Prolonged AV conduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right ventricular stimulation (Active Comparator): patients with conventional Right Ventricular Stimulation (only RV) with optimized algorithms for minimization of pacing
  Interventions: Device: Dual chamber pacemaker
- Biventricular Stimulation (Experimental): Patients with biventricular stimulation (Right Ventricle and Left Ventricle)
  Interventions: Device: Cardiac resynchronization therapy pacemaker

INTERVENTIONS:
Device: Cardiac resynchronization therapy pacemaker — biventricular stimulation with cardiac resynchronization therapy pacemaker (crt-p)
  Arms: Biventricular Stimulation
Device: Dual chamber pacemaker — right ventricular stimulation with dual chamber pacemaker
  Arms: Right ventricular stimulation

SUMMARY:
This study was designed to evaluate the potential benefits of treatment with biventricular device in patients with normal systolic function , indication for pacing and impaired atrio-ventricular conduction , by comparing the treatment with dual-chamber device . The REAL -CRT study is designed to test the hypothesis that, in patients with atrioventricular block of I degree and standard pacing indications , biventricular pacing is superior to single stimulation of the right ventricle (RV) with optimized algorithms for minimization of pacing , as assessed by echocardiography an endpoint defined in terms of maintenance over time of left ventricular ejection fraction (LVEF ) and left ventricular end-systolic volume ( LVESV ) .

DETAILED DESCRIPTION:
Clinical data suggest that biventricular pacing is able to preserve the myocardial performance more effectively than the right ventricular pacing in patients with atrioventricular block and mild systolic dysfunction . In particular, some studies have shown that medical therapy in these patients could be responsible for an increase in the cumulative percentage of chronic pacing over the 40% threshold , the threshold associated with a higher incidence of atrial fibrillation and hospitalization for heart failure and ventricular arrhythmias . In addition , patients with pre-existing left ventricular dysfunction and indication for pacing standards have improved left ventricular systolic function , exercise capacity and quality of life as a result of biventricular pacing as compared with Right ventricular pacing . These results suggest that biventricular pacing is a feasible option for permanent pacing in patients who have normal systolic function of the left ventricle and that this can be altered from the adverse effects of conventional Right ventricular pacing on systolic function of the left ventricle . This reality has prompted physicians to assess the value and role of cardiac resynchronization therapy (CRT ) in patients with prolonged Atrio-Ventricular (AV) conduction . Note the deleterious effects of chronic stimulation of the right ventricle , the optimal pacing mode should always be considered in these patients at the time of implantation . This study was designed to evaluate the potential benefits of treatment with biventricular device in patients with normal systolic function , indication for pacing and impaired atrio-ventricular conduction, by comparing it with the treatment with dual chamber device

ELIGIBILITY:
Inclusion Criteria:

* Patients with standard indications to stimulation with a high probability of paced beats according to the clinical evaluation of the investigators:
* First degree AV block (PR ≥ 220 ms) and indication for pacing
* Paroxysmal AV block second degree (Type I and Type II) associated with long-PR (PR ≥ 220 ms)
* Patient must be able to attend all required follow-up visits at the study center.
* LVEF> 35%

Exclusion Criteria :

* Patient is less than 18 years of age.
* Patients with a life expectancy less than 12 months
* Indication for CRT in class I and II
* Third-degree AV block
* Patients currently enrolled in other studies / logs
* Patients who are not able to understand and sign an informed consent
* State of current or planned pregnancy within 12 months of enrollment
* Inability to understand and complete the questionnaire QOL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
LVEF | 2 years
  LVEF (Left Ventricular Ejection Fraction: such as the assessment of systolic function of the left ventricle)
LVESV | 2 years
  LVESV (Left Ventricular End Systolic Volume: such as the assessment of left ventricular remodeling)

SECONDARY OUTCOMES:
echocardiographic left ventricular measures | 2 years
  . Structure and cardiac function:
  * Left ventricular End Systolic Diameter, Left ventricular End Diastolic Diameter
  * Left Ventricular End Systolic
Echocardiographic altrial measures | 2 years
  Size of the left atrium (diameter and volume)
Clinical outcome | 2 years
  Clinical benefit:
  * 6 minute walking test
  * quality of life questionnaire
  * New York Heart Association class
  * number and duration of hospitalizations
Atrial fibrillation (AF) | 2 years
  Incidence of AF:
  * incidence of persistent AF
  * burden of FA
  * new onset of AF

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Botto, Principal Investigator — S. Anna Hospital
Locations (1):
- Azienda Ospedaliera Sant'Anna, Como, Como, Italy

REFERENCES:
- [Derived] Botto GL, Iuliano A, Occhetta E, Belotti G, Russo G, Campari M, Valsecchi S, Stabile G. A randomized controlled trial of cardiac resynchronization therapy in patients with prolonged atrioventricular interval: the REAL-CRT pilot study. Europace. 2020 Feb 1;22(2):299-305. doi: 10.1093/europace/euz321. PMID 31722381